CLINICAL TRIAL: NCT03771781
Title: A Single-Center, Open-Label, Randomized, Single-Dose, Two-Period, Two-Sequence, Crossover Study to Assess the Bioequivalence of Test Formulation With Reference Formulation in Healthy Adult Subjects.
Brief Title: Bioequivalence Study of Empagliflozin Tablet in Healthy Participants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTTQ-BE-2018-EGLJ
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin Tablets (Other): The test formulation is manufactured by Jiangsu Chia-tai Tianqing Pharmaceutical Co.,Ltd.During the study session,subjects will be administered a single does of Empagliflozin Tablets 25mg after fasting and fed conditions.
  Interventions: Drug: Empagliflozin Tablets
- Empagliflozin Tab 25 MG (Other): The reference formulation is manufactured by Boehringer Ingelheim International GmbH.During the study session,subjects will be administered a single does of Empagliflozin Tab 25 MG after fasting and fed conditions.
  Interventions: Drug: Empagliflozin Tab 25 MG

INTERVENTIONS:
Drug: Empagliflozin Tablets — Observe the safty and PK after subjects receiving a single dose of Empagliflozin Tablets.
  Arms: Empagliflozin Tablets
Drug: Empagliflozin Tab 25 MG — Observe the safty and PK after subjects receiving a single dose of Empagliflozin Tablets( Jardiance®）.
  Arms: Empagliflozin Tab 25 MG

SUMMARY:
Bioequivalence Study of Empagliflozin Tablets and Jardiance® Under Fasting and Fed Conditions in Chinese Healthy Volunteers.

DETAILED DESCRIPTION:
A Single-Center,Open-Label,Randomized,Single-Dose,Two-Period,Two-Sequence,Crossover Study to Assess the Bioequivalence of Test Formulation Empagliflozin Tablets with Reference Formulation Jardiance® in Chinese Healthy Adult Subjects under Fasting and Fed Conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 50 years, inclusive.
2. The body weight of male is not less than 50kg, and female is not less than 45kg. All participants' body mass index (BMI) is between 19~26.
3. Subjects are fully informed and voluntarily consent to participate in this study.
4. Volunteers can communicate well with researchers and comply with the requirements of this study.

Exclusion Criteria:

1. Any with chronic or active gastrointestinal diseases such as esophageal diseases, gastritis, gastric ulcers, enteritis, active gastrointestinal bleeding or got any digestive tract surgery within three years.
2. Any disease previously or currently suffering from circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry, and metabolic abnormalities, and which the researchers believe can interfere with the results of the test.
3. Any history of allergy to drugs, food, or other substances.
4. Dysphagia, difficulty in collecting blood or halo needle, history of dizziness.
5. Those who have undergone surgery during the first four weeks of the trial or are scheduled to perform surgery during the study period.
6. Those who has taken any drug (including vitamin products, Chinese herbs) within 14 days before the study.
7. Those who use any inhibits or induces hepatic metabolism within 30 days before the study.
8. Those who participated in any clinical drug trial within 3 months prior to the trial.
9. Those who donated or lose massive blood within 3 months before the study (> 450 ml).
10. Pregnant and lactating women.
11. Male subjects (or their partners) or female subjects had unprotected sex or pregnancy plans within 2 weeks before screening and 6 months after the end of the trial, Those who are unwilling to use one or more non-drug contraceptive methods (e. G. Complete abstinence, contraceptive ring, partner ligation, etc.) during the study.
12. Drug abusers or those who have used soft drugs for 3 months before the trial or who took hard drugs one year before the study.
13. Those who has special requirements for diet and is unable to follow a uniform diet.
14. Smokers or those who smoked more than 5 cigarettes a day 3 months before the study.
15. An alcoholic or regular drinker for six months before the study, that is, a person who drinks more than 14 units of alcohol a week.
16. People who drink excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250 mL) per day or who do not agree to stop drinking tea, coffee and/or caffeinated beverages during the study period.
17. Those who take drug or food which may affect the drug metabolism(including grapefruit or grapefruit products, dragon fruit, mango, pomelo, orange, yellow purine diet).Or the researchers think that there are other affect drug absorption, distribution, metabolism and excretion of diet.Or refuse to stop eating the diet during the study.
18. Those with abnormal physical examination, electrocardiogram, laboratory examination, vital signs and test related examination with clinical significance .
19. Those who has vital signs with clinical significance, positive urine screening test, positive alcohol breath test or positive female urine pregnancy.
20. Those who has acute illness or concomitant medication occurred before participating in the study.
21. Other reasons which,in the opinion of the medical investigator,would prevent the subject from participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0hours、0.67hours、1hours、1.5hours、2hours、2.5hours、3hours、4hours、6hours、8hours、12hours、24hours、36hours、48hours、72hours
  Maximum observed plasma concentration following drug administration from the raw plasma concentration-time data.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curves (AUC) | 0hours、0.67hours、1hours、1.5hours、2hours、2.5hours、3hours、4hours、6hours、8hours、12hours、24hours、36hours、48hours、72hours
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China